CLINICAL TRIAL: NCT04349332
Title: Early Extubation for Patients With Acute Hypoxemic Respiratory Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was not initiated, no subjects enrolled.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB20-0594
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Mechanical Ventilation; Corona Virus Infection
Keywords: helmet interface NIV; early extubation; acute hypoxemic respiratory failure
MeSH Terms: conditions — Coronavirus Infections; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Helmet non invasive ventilation (NIV) (Active Comparator): Patients randomized to the intervention group will be extubated to helmet NIV.
  Interventions: Device: Helmet non-invasive ventilation (NIV)
- Control invasive mechanical ventilation (No Intervention): Patients randomized to the control group will continue invasive mechanical ventilation. Once weaning criteria are met, patients will undergo a spontaneous breathing trial for 30 minutes. If the spontaneous breathing trial is successful, then the patient will be extubated.

INTERVENTIONS:
Device: Helmet non-invasive ventilation (NIV) — After application of the helmet, arterial blood gas sampling will be utilized to follow gas-exchange; Noninvasive support will be reduced progressively in accordance to clinical improvement and will be discontinued if patient maintains respiratory rate <30breaths/min and PaO2 >75mm Hg with FiO2 0.5 without ventilatory support. If endotracheal intubation is required, the helmet will be removed and the patient will be intubated without delay.
  Arms: Helmet non invasive ventilation (NIV)

SUMMARY:
The objective of the study is to evaluate the efficacy of helmet NIV in reducing the duration of invasive mechanical ventilation in order to minimize ventilator needs during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Single center randomized clinical trial investigating the efficacy of helmet NIV used for early liberation from mechanical ventilation in patients with acute hypoxemic respiratory failure.

Intervention: Helmet group Patients randomized to the intervention group will be extubated to helmet NIV without a spontaneous breathing trial. The helmet will be connected to oxygen and room air flow meter to deliver a minimum of 60L of fresh gas flow and a PEEP valve. The PEEP will be increased using a PEEP valve in increments of 2-3 cmH20 to improve peripheral oxygen saturation of at least 90% at an inspired oxygen requirement (FiO2) of ≤ 60%.14 After application of the helmet, arterial blood gas sampling will be utilized to follow gas-exchange; this is a part of usual care for the management of patients with acute hypoxemic respiratory failure. Noninvasive support will be reduced progressively in accordance to clinical improvement and will be discontinued if patient maintains respiratory rate <30breaths/min and PaO2 >75mm Hg with FiO2 0.5 without ventilatory support. If endotracheal intubation is required, the helmet will be removed and the patient will be intubated without delay.

Control: Usual Care Patient randomized to the control group will continue invasive mechanical ventilation until the following weaning criteria are met:15 Resolution or improvement of the condition leading to intubation Hemodynamic stability, defined as systolic blood pressure between 90 and 160 mm Hg and heart rate less than 140/min without vasopressors or with low doses of vasopressors Glasgow Coma Scale score of 13 or greater Respiratory stability (oxygen saturation >90% with fraction of inspired oxygen [Fio2] ≤0.4, respiratory rate <35/min, Noncopious secretions (<3 aspirations in the last 8 hours).

Once weaning criteria are met, patients will undergo a spontaneous breathing trial for 30 minutes on pressure support mode. Criteria for failure to tolerate the SBT were agitation, anxiety, low level of consciousness (Glasgow Coma Scale score <13), respiratory rate higher than 35/min and/or use of accessory muscles, oxygen saturation by pulse oximetry less than 90% with Fio2 higher than 0.5, heart rate higher than 140/min or greater than a 20% increase from baseline, systolic blood pressure lower than 90 mm Hg, or development of arrhythmia. If the spontaneous breathing trial is successful, then the patient will be extubated.

Subjects will be followed for long term followup at 90 day and 1year mortality

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years old on mechanical ventilation for at least 48 hours Positive End Expiratory Pressure (PEEP) level between 8 to 13cm H20 The ratio between the partial pressure of oxygen and fraction of inspired oxygen (PaO2/FiO2) between 150 and 300 mmHg with FiO2≤0.6 pH≥7.25 Respiratory rate (RR)≤30/min Adequate gag and cough reflex Ability to spontaneously breathe

Exclusion Criteria:

Hemodynamic instability (Systolic blood pressure <90 or requiring >2 vasoactive agents) Tracheostomy Upper airway obstruction Pregnancy Elevated intracranial pressure Upper airway obstruction Glasgow coma scale ≤ 8 Patients who refuse to undergo endotracheal intubation, whatever the initial therapeutic approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-01-09 (Estimated); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
ventilator days | up to 4 weeks
  duration of mechanical ventilation via endotracheal tube

SECONDARY OUTCOMES:
Intensive care unit (ICU) length of stay | up to 6 weeks
  number of days admitted to the ICU
need for re-intubation | up to 6 weeks
  number of patients requiring endotracheal intubation after extubation

OTHER OUTCOMES:
hospital length of stay | up to 6 weeks
  number of days spent in hospital during enrollment hospitalization
hospital mortality | up to 6 weeks
  death from any cause during hospitalization time of enrollment
long term mortality | up to 1 year
  death from any cause 90 day, 1year
ICU related complications | up to 6 weeks
  including ventilator associated pneumonia, GI hemorrhage, DVT/PE, sacral decubitus ulcer, delirium, ICU acquired weakness
discharge location | up to 90 days
  measure the location (home, rehabilitation center, nursing home)
health care utilization | up to 6 weeks
  days alive and institution free
diaphragm ultrasound thickness | up to 6 weeks
  ultrasound measurement at end expiration: enrollment, pre extubation, post extubation
diaphragm thickening fraction | up to 6 weeks
  ultrasound measurement at end expiration and inspiration to calculate thickening fraction

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No